CLINICAL TRIAL: NCT06151535
Title: An Open-label Study Evaluating the Safety and Effectiveness of Intradermal Injections of ELAPR002f Injectable Gel in the Improvement of Multiple Attributes of Skin Quality in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Effectiveness of ELAPR002f Injectable Gel for the Improvement of Skin Quality in Adult Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2028-601-008
Record Dates: First submitted 2023-11-22; First posted 2023-11-30 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Skin Quality Deficit
Keywords: Skin Quality Deficit; ELAPR002f Injectable Gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ELAPR002f Injectable Gel (Experimental): Participants will receive 3 treatment sessions 1 month apart of ELAPR002f injectable gel and will be followed for 4 months.
  Interventions: Device: ELAPR002f Injectable Gel

INTERVENTIONS:
Device: ELAPR002f Injectable Gel — Intradermal Injections

SUMMARY:
Elastin is a protein found in the dermis of the skin that is gradually lost with aging which impacts skin tissue and leads to reduced structural integrity, hydration, and elasticity of the skin, resulting in loose skin and the formation of folds and wrinkles. Loose skin, folds, and wrinkles can be treated by injecting biocompatible structures to fill the the affected area and improve elasticity/hydration upon implantation. The purpose of this study is to evaluate the safety and effectiveness of ELAPR002f injectable gel in adult participants for the improvement of skin quality in adults.

ELAPR002f injectable gel is an investigational device being developed for the improvement of facial skin quality attributes such as fine lines, elasticity, and hydration. Approximately 30 participants 30 to 60 years of age seeking improvement of skin quality will be enrolled.

Participants will receive 3 treatment sessions, 1 month apart, of ELAPR002f injectable gel to each cheek and behind 1 ear (for histological assessment) and will be followed up for up to 4 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants in general good health, in the opinion of the investigator, with no known active COVID-19 infection, seeking improvement of facial skin quality.
* Moderate or severe (symmetric grade 2 or 3 on the Allergan Fine Lines Scale [AFLS] and Allergan Cheek Smoothness Scale [ACSS]) fine lines and cheek smoothness scores on both cheeks based on investigator's live assessment.
* Each cheek is amenable to at least a 1 point improvement on the AFLS and ACSS.

Exclusion Criteria:

* Current cutaneous or mucosal inflammatory or infectious processes (eg, herpes), rosacea, abscess, an unhealed wound, active acne, or a cancerous or precancerous lesion, on the face or behind the ears.
* History of pigmentation disorders or current pigmentation disorder on the face or behind the ears.
* Active smoker.
* Currently using topical retinoids, or have used topical retinoids in the past 60 days (2 months) on the face or behind the ears.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Responder Status Based on Evaluating Investigator's Live Assessment of Each Cheek Separately Using Allergan Cheek Smoothness Scale (ACSS) | Up to 8 months
  The ACSS is a 5-point photonumeric scale that assesses the appearance of cheek smoothness vs coarseness where 0=none and 4=extreme. A responder is a participant with at least 1-grade improvement from baseline in ACSS.
Percentage of Participants Achieving Responder Status Based on Evaluating Investigator's Live Assessment of Each Cheek Using Allergan Fine Line Scale (AFLS) | Up to 8 months
  The AFLS is a 5-point photonumeric scale that assesses the appearance of fine lines where 0=none and 4=diffuse superficial lines. A responder is a participant with at least 1-grade improvement from baseline in AFLS.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- CRC - Centro Ricerche Cliniche di Verona S.r.l. /ID# 226370, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=2028-601-008